CLINICAL TRIAL: NCT04110483
Title: Safety and Short-term Oncological Outcomes of Thulium Fiber Laser En-bloc Resection of Non-muscle-invasive Bladder Cancer
Brief Title: Thulium Fiber Laser En-bloc Resection vs Conventional Transurethral Resection of Non-muscle-invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sechenov-ERBT-16
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TURBT (Active Comparator): A step-by-step resection of a tumor. Firstly, visible tumor is resected, then resection continues to the apparently normal mucosa on the border of the tumor, than resection of the muscle layer at the base of the tumor is performed until normal muscle fibers are visible.
  Interventions: Procedure: Transurethral resection of non-muscle-invasive bladder cancer
- Tm-fiber ERBT (Experimental): A circumferential incision around the tumor is made in the visually intact bladder mucosa. After that, the incision is continued deeper into the muscular layer. Than the surgeon resects the base of the tumor with the muscular layer using traction and incisions of the muscle fibers.
  Interventions: Procedure: Thulium fiber laser en-bloc resection of non-muscle-invasive bladder cancer

INTERVENTIONS:
Procedure: Thulium fiber laser en-bloc resection of non-muscle-invasive bladder cancer — After cystoscopy and determining tumor topography, a circumferential incision around the tumor is made in the visually intact bladder mucosa (approximately 10 mm from the edges of the tumor). It allows for accurate morphological evaluation of the surgical margin. After that, the incision is continued deeper into the muscular layer. Having identified the layer, the surgeon resects the base of the tumor with the muscular layer using traction and incisions of the muscle fibers. Making incisions in the muscular layer requires precision, a full bladder and adequate guidance with visualization techniques. Traction may be employed with the help of the tip of the resectoscope or working element. After complete tumor resection, local hemostasis was performed.
  Arms: Tm-fiber ERBT
Procedure: Transurethral resection of non-muscle-invasive bladder cancer — After cystoscopy and determining tumor topography, a step-by-step resection of a tumor is done. Firstly, visible tumor is resected, then resection continues to the apparently normal mucosa on the border of the tumor, than resection of the muscle layer at the base of the tumor is performed until normal muscle fibers are visible.
  Arms: TURBT

SUMMARY:
Ongoing efforts aim at overcoming the challenges of conventional transurethral resection of bladder tumor (TURBT) such as the high recurrence rate, difficulty of pathologic interpretation and complications including wall injury. Possible advantages may have en bloc resection of bladder tumor which was previously shown to be effective and safe technique. Use of novel thulium-fiber laser may also provide additional safety and efficacy of the resection.

Objective. To prospective assess the safety and efficacy of Thulium-fiber en bloc resection of bladder tumor (Tm-fiber-ERBT) compared to TURBT.

DETAILED DESCRIPTION:
En bloc resection of bladder tumor (ERBT) was first employed by Kawada T. et al. in 1997. The technique showed promising results in terms of safety and tumor staging. Development of laser surgery and emergence of the holmium (Ho:YAG) and later thulium (Tm:YAG) lasers in the 1990s enabled laser ERBT with subsequent studies demonstrating high efficacy and safety of the new techniques. Ho:YAG and Tm:YAG ERBT have distinct advantages over conventional TURBT such as the complete absence of the obturator nerve reflex and hence, lower risks of perforation or bleeding as well as a higher quality specimens for pathologic examination, due to lack of the cautery effect. Recently, a new type of thulium laser was developed - that allows to decrease the penetration depth less than 0.15 mm, which is two times less than that of Tm:YAG. Another advantage is the decreased carbonization compared to Tm:YAG due to better water absorption of laser energy. All these aspects make Tm:YAG a precise tool that may improve the resection quality resulting in better management. Data on laser ERBT of NMIBC with Tm:YAG is limited and that on Tm-fiber laser ERBT is absent altogether. The investigators hypothesized that Tm-fiber laser ERBT would result in a lower probability of adverse events and better recurrence-free survival compared to conventional TURBT.

ELIGIBILITY:
Inclusion Criteria:

• Primary Ta or T1 bladder cancer (NMIBC)

Exclusion Criteria:

• Pure carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival rate | 3 month
  Absence of cancer at the site of previous resection on histological examination after re-biopsy

SECONDARY OUTCOMES:
Detrusor presence in the specimen | 1 day after the surgery
  The presence of muscle fibers in specimens on histological investigation
Complications | up to 1 year
  Rate of postoperative complications, their severity according Clavien-Dindo score

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, M.D., Ph.D., Principal Investigator — Sechenov University
Locations (1):
- Clinic of Urology, Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No